CLINICAL TRIAL: NCT06961890
Title: Change in Hygiene and Sugar Comsuption Habits After Use of Cognitive Behavioral Therapy in Pediatric Dentistry in Twins
Acronym: CARDEC-BC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Mariana Minatel Braga, Phd, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARDEC-TWINS-BC
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Oral Manifestations; Child Behavior; Adolescent Behavior; Change; Cognitive
Keywords: clinical study; cognitive behavioral therapy; oral health; twins; motivational guidance; preference patients
MeSH Terms: conditions — Oral Manifestations; Child Behavior; Adolescent Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cognitive behavioral therapy (Experimental): All participants will receive a standardized orientation for changing oral health habits using principals of cognitive behavioral therapy
  Interventions: Behavioral: Principals of cognitive behavioral therapy on guided changing hygiene and sugar comsuption habits

INTERVENTIONS:
Behavioral: Principals of cognitive behavioral therapy on guided changing hygiene and sugar comsuption habits — The twin pairs will also receive guidance on healthy sugar consumption and oral hygiene habits, as the first intervention among the dental interventions received. For the baseline assessment, each participant answered a questionnaire about their diet the day before and about oral hygiene, in addition to demonstrating how they perform it. Thus, the cognitive behavioral theory was applied, so that the participant can record the goals achieved weekly and monthly.

SUMMARY:
The objective of this study is to verify the changing habits and their maintenance after using cognitive behavioral therapy, exploring factors that may be associated with these stages and the moment in which they occur.

DETAILED DESCRIPTION:
The objective of this clinical trial is to verify the time until changing habits and their maintenance after using cognitive behavioral therapy, exploring the following factors that may be associated with these stages and the moment in which they occur:

* Evaluate the cost-effectiveness of guidance based on cognitive behavioral therapy in relation to changes aimed at oral hygiene and diet habits, through a before and after study;
* Investigate individual and contextual preferences associated with adherence and maintenance of behaviors associated with oral health (diet and oral hygiene) through a Discrete Choice Experiment (DCE)
* Measure the effect of retaining hygiene and diet guidance on pairs who did not submit the calendar and on those who submitted the calendar.

ELIGIBILITY:
Inclusion Criteria:

* Twin children born at the Hospital de Clínicas de São Paulo between 2007 and 2014;
* Children whose mothers were followed up at the Multiple Pregnancy Unit;
* Guardians who sign the informed consent form;
* Children who sign the assent form.

Exclusion Criteria:

* Children whose families that cannot be contacted by phone call, email, or social media;
* Children with medical or psychological conditions that prevent safe participation in the dental research.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2028-08-02 (Estimated)

PRIMARY OUTCOMES:
Changing hygiene habits and sugar consumption in children and adolescents | 6 months
  Assessed using a 12-point checklist performed at baseline and at 6 month follow-ups

SECONDARY OUTCOMES:
Preference for attributes associated with adherence to oral health-related behavior | 24 months
  It will be measured after 12 months of the intervention (guidance and motivation) applied to the twins through a Discrete Choice Experiment
Maintenance hygiene habits and sugar consumption in children and adolescents | 12, 18, 24 months
  Assessed using a 12-point checklist performed at baseline and at 12, 18 and 24 month follow-ups, in which it will be assessed whether there was improvement, worsening or return to initial conditions.

OTHER OUTCOMES:
Costs associated with the initial intervention that resulted in the effect of habit change | 24 months
  For the costs, the direct and indirect costs necessary for the intervention carried out at baseline and at the 6, 12, 18 and 24 month follow-ups were considered
Visual attention metrics | 24 months
  Examples of metrics evaluated will be viewing time, fixations, saccades, among others, which will be measured by the eye-tracking device, during the use of images, videos and demonstrations in models during the evaluation process. Visual reports such as gaze plots (gaze plots) and heat maps (areas of greatest gaze fixation - heatmaps) will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, Principal Investigator — University of Sao Paulo; Edgard M Crosato, Study Director — University of Sao Paulo; Thais GO Machado, Study Chair — University of Sao Paulo; Fausto M Mendes, Study Director — University of Sao Paulo; Laura RA Pontes, Study Chair — University of Sao Paulo
Locations (1):
- Faculdade de Odontologia da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected on pregnancy, parental sociodemographics (age, sex), alloparental care, and twin characteristics (age, sex, zygosity), using questionnaires and registry data (birth weight, ICU admission, chorionicity, gestational age, fetal growth, complications). Caries lesions and indicators of physical, cognitive, and emotional development will be monitored. Behavioral and physiological data will be collected before and during a dental procedure. Instruments include the Danish Twin Registry Zygosity Questionnaire, Environmental Sensitivity, Socialization Goals, Alabama Parenting, Twin Relationship, Childhood Adversity, Quality of Life, MCDAS-f, Emotion Regulation Checklist, and identity fusion. Additional data: caries detection (ICDAS), physical (height, weight), cognitive (Raven), figure drawings, videos, facial temperature (thermal camera), voice recordings, and saliva swabs. Metadata will follow USP's Open Access Policy, including DOI, title, authors, and deposit details.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: baseline, 6M, 12M, 18M, 24M
Access Criteria: Data will be collected on pregnancy, parental sociodemographics (age, sex), alloparental care, and twin characteristics (age, sex, zygosity), using questionnaires and registry data (birth weight, ICU stay, chorionicity, gestational age, fetal growth, complications). Caries lesions and indicators of physical, cognitive, and emotional development will be monitored. Behavioral and physiological data will be gathered before and during dental procedures. Instruments include Zygosity Questionnaire, Environmental Sensitivity, Socialization Goals, Alabama Parenting, Twin Relationship, Childhood Adversity, Quality of Life, MCDAS-f, Emotion Regulation, and identity fusion. Additional data: caries detection (ICDAS), physical (height, weight), cognitive (Raven), figure drawings, videos, facial temperature (thermal camera), voice recordings, and saliva swabs. Metadata will follow USP Open Access Policy with DOI, title, authors, keywords, funding, and deposit info.